CLINICAL TRIAL: NCT01203449
Title: Development of Standards for the New Ballard Maturation Score
Acronym: Ballard
Status: Completed | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Edward F. Donovan/ Lead Principal Investigator, Cincinnati Children's Medical Center
Other Study IDs: NICHD-NRN-0012; U10HD027853 (NIH); U10HD027871 (NIH); U10HD021385 (NIH); U10HD027880 (NIH); U01HD019897 (NIH); U10HD021364 (NIH); U10HD021415 (NIH); U10HD027851 (NIH); U10HD021373 (NIH); U10HD027856 (NIH); U10HD027881 (NIH); M01RR008084 (NIH); M01RR006022 (NIH); M01RR000750 (NIH); M01RR000070 (NIH); M01RR000997 (NIH); U10HD021397 (NIH)
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Pregnancy
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Prematurity; Gestational Age
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of this study was to evaluate the accuracy of gestational age (GA) estimates by using the New Ballard Score (NBS) in newborns 24 to 27 weeks GA with accurate obstetric estimates of GA. Secondary purposes were: (1) to compare the accuracy of GA estimates derived from the NBS, the original Ballard score, and the physical items of the original Ballard score and (2) to compare these measures of GA and best obstetric estimates of GA as predictors of survival, morbidity, and hospital stay among infants <28 weeks' gestation and among very low birth weight infants in general.

DETAILED DESCRIPTION:
The Ballard maturational assessment is commonly used to estimate gestational age (GA) when the menstrual history and other obstetrical estimates of GA are uncertain. The original Ballard Score and the New Ballard Score are based on the assumption that the fetal skin, subcutaneous tissues, and neuromuscular system mature at predictable rates.

Because of variation in maturation rates among healthy fetuses or abnormalities of fetal development, fetal maturation can vary at a given GA. For very premature infants, small differences in GA result in large differences in outcome and may even determine whether intensive care is given.

The primary purpose of this study was to evaluate the accuracy of GA estimates by using the NBS in newborns 24 to 27 weeks GA with accurate obstetric estimates of GA. Secondary purposes were: (1) to compare the accuracy of GA estimates derived from the NBS, the original Ballard score, and the physical items of the original Ballard score and (2) to compare these measures of GA and best obstetric estimates of GA as predictors of survival, morbidity, and hospital stay among infants <28 weeks' gestation and among very low birth weight infants in general.

For this study, eligible infants included those with birth weights of 401-1500g born in the National Institute of Child and Human Development (NICHD) Neonatal Research Network (NRN). Before 48 hours of age, enrolled infants were examined using the New Ballard Score by trained and certified research nurses masked to obstetric estimates of gestational age. A best obstetrical estimate of GA, used for screening of potentially eligible infants, was determined from the last menstrual period, obstetrical measures, and ultrasound findings recorded on the labor and delivery records.

ELIGIBILITY:
Inclusion Criteria:

* <28 weeks gestational age by best obstetrical estimate
* Availability of mother's prenatal records for review
* First prenatal visit occurred before 17 weeks' gestation
* Mother's menstrual history allowed calculation of GA at birth
* Mother reported the duration of her usual menstrual cycles as 21 to 35 days
* Mother had 3 consecutive normal menstrual cycles before the missed menstrual period identifying the index pregnancy
* Mother reported that she was certain within 4 days of the first day of the last menstrual period (as recorded at the time of the first prenatal visit)
* Mother denied use of birth control medication during the 3 months preceding the last menstrual period.

Exclusion Criteria:

* Inaccurate or unavailable menstrual histories

Max Age: 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants born in the NICHD Neonatal Research Network during the study period.
Sampling Method: Probability Sample
Enrollment: 1090 (Actual)
Dates: Start 1994-06; Primary Completion 1996-03 (Actual); Study Completion 1996-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward F. Donovan, MD, Study Director — Children's Hospital Medical Center, Cincinnati; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; Seetha Shankaran, MD, Principal Investigator — Wayne State University; David K. Stevenson, MD, Principal Investigator — Stanford University; Raymond Bain, PhD, Principal Investigator — George Washington University; Avroy A. Fanaroff, MD, Principal Investigator — Case Western Reserve University; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee at Memphis; Barbara J. Stoll, MD, Principal Investigator — Emory University; Jon E. Tyson, MD MPH, Principal Investigator — University of Texas; James A. Lemons, MD, Principal Investigator — Indiana University; Lu-Ann Papile, MD, Principal Investigator — University of New Mexico
Locations (11):
- United States (11):
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Result] Donovan EF, Tyson JE, Ehrenkranz RA, Verter J, Wright LL, Korones SB, Bauer CR, Shankaran S, Stoll BJ, Fanaroff AA, Oh W, Lemons JA, Stevenson DK, Papile LA. Inaccuracy of Ballard scores before 28 weeks' gestation. National Institute of Child Health and Human Development Neonatal Research Network. J Pediatr. 1999 Aug;135(2 Pt 1):147-52. doi: 10.1016/s0022-3476(99)70015-6. PMID 10431107
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/